CLINICAL TRIAL: NCT00741546
Title: Association of Low Vitamin D Levels With Mortality in Patients With Reduced Left Ventricular Function Referred to Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Dr.med. F. Bakhtiary, Depratment of Thoracic and Cardiovascular Surgery
Other Study IDs: Vitamin D in cardiac surgery
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2008-08-26 (Estimated); Status verified 2008-08

CONDITIONS: Malnutrition
Keywords: Vitamin D; malnutrition; cardiac surgery; study; emphasize; importance; significant; high risk patient
MeSH Terms: conditions — Malnutrition | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A: Patients referred for cardiac surgery intervention
  Interventions: Procedure: Cardiac Surgery

INTERVENTIONS:
Procedure: Cardiac Surgery — Cardiac Surgery

SUMMARY:
This study investigates if reduced serum levels of vitamin D concentration are a typical feature in patient group with low left ventricular function admitted for cardiac surgery interventions. and also the necessity of more preventive strategies for adequate nutrition of these patients with more focus on intake of vitamin D before admission to cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* All routinely cardiac procedures

Exclusion Criteria:

* dialysis, cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted for cardiac surgery intervention
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2007-03; Primary Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Perioperative mortality | 90day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Thoracic and Cardiovascular Surgery, Frankfurt am Main, Hesse, Germany